CLINICAL TRIAL: NCT00159484
Title: Phase I/II Study of Celebrex and EPO906 in Patients With Metastatic Colorectal Cancer (CEPO906AUS10)
Brief Title: Phase I/II Study of Celebrex and EPO906 in Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3c-03-19
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Colon Cancer; Colorectal Cancer
Keywords: phase 1; phase one; phase I
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — epothilone B; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): EPO906, celecoxib
  Interventions: Drug: EPO906, celecoxib

INTERVENTIONS:
Drug: EPO906, celecoxib — EPO906 IV, every three weeks, celecoxib by mouth twice a day every day

SUMMARY:
This study is for people with advanced colorectal cancer. This study uses the drugs Celebrex and EPO906. EPO906 is an experimental drug that has not been approved by the FDA. EPO906 is a drug that has been shown in the laboratory to cause cancer cells to die and prevents them from growing and reproducing. Celebrex is a drug that is approved by the FDA for the treatment of arthritis and prevention of colon polyps. Colon polyps are small growths in the colon. If not surgically removed, some colon polyps can become cancerous. Some studies have shown that Celebrex may reduce the side effects of chemotherapy. Other studies have shown that it may increase the effectiveness of some chemotherapy. Celebrex is not approved by the FDA for reducing the side effects of chemotherapy or improving the effectiveness of chemotherapy. The combination of EPO906 and Celebrex in this study is experimental.

The main goal of this study is to see if adding the drug Celebrex to the drug EPO906 will decrease the amount of diarrhea seen in patients that receive EPO906.

The goal of the first phase of this study is to find the highest dose of EPO906 that can be given safely with Celebrex. The dose of Celebrex will remain the same for the whole study. Higher doses of EPO906 will be given to each group of patients. The increase of EPO906 will stop once more than one patient has serious side effects. The highest dose of EPO906 that can be given with Celebrex (without serious side effects) will be called the pilot dose.

The goal of the second phase of this study is to find out how tumors respond to these doses of the drugs. Another purpose of this study is to see how the body processes the EPO906 and Celebrex. This study will also look at the side effects of these drugs. In this study, we will measure how long subjects live, how often tumors shrink after receiving the study drugs, and how long it takes for tumors to increase in size after receiving the study drugs. This study will also measure the levels of genes, which are the cell's blueprint, in participant's tumors. Several genes can affect how people's bodies react to the cancer drugs. Genes will also be measured in participant's blood. We want to see if these predict response to the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the colon or rectum for which no further standard chemotherapy is considered to be effective. Patients must have failed 5-FU, CPT-11 and/or oxaliplatin based chemotherapy.
* SWOG performance status 0-1
* ANC>1000, platelets >100,000.
* Total bilirubin < 2 x upper limit of normal. Transaminase (AST and/or ALT) < 2 x upper limit of normal or < 5 x upper limit of normal in patients with liver metastasis.
* Serum creatinine < 1.25 x institutional upper limit of normal.
* Female patients of child-bearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing.

Exclusion Criteria:

* Patient has received any other investigational agent within 28 days of first day of study drug dosing.
* History of another malignancy within 3 years prior to study entry, except curatively treated non-melanoma skin cancer, prostate cancer, or cervical cancer in situ.
* Patient has another severe and/or life-threatening medical disease.
* Patient has an acute or known chronic liver or kidney disease (e.g., chronic active hepatitis, cirrhosis, chronic renal insufficiency).
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient has received chemotherapy within 4 weeks (6 weeks for nitrosourea, mitomycin-C or any antibody therapy)
* Patients with symptomatic brain metastasis.
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria. (e.g. congestive heart failure, myocardial infarction within 6 months of study)
* Medical, social or psychological factors interfering with compliance.
* Patients who have undergone major surgery for any cause less than 4 weeks prior to study entry.
* Patients taking Coumadin® or other agents containing warfarin, with the exception of low dose Coumadin® (1 mg or less) administered prophylactically for maintenance of in-dwelling lines or ports.
* Any peripheral neuropathy > Grade 1.
* Patients with unresolved diarrhea > Grade 1.
* Patients may not have a history of an allergy to sulfonamide drugs.
* Patients may not have active peptic ulcer disease or other contraindications to chronic NSAID use or aspirin use.
* Patients with lactose intolerance.
* Patients taking full-dose NSAIDs, including aspirin, regularly for any reason (e.g., arthritis,history of TIA or myocardial infarction). Patients taking cardiac preventive dose ASA (<81mg daily) are eligible. Patients should stop taking any other NSAIDs 14 days prior to receiving first dose of Celecoxib.
* Patients with hypersensitivity to COX-2 inhibitors, NSAIDS or salycilate.
* Patients taking fluconazole or lithium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-10; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of Celebrex in combination with EPO906 in patients with metastatic colorectal cancer. | One month
Once MTD is established we propose to expand the dose level of the MTD to 62 new patients to evaluate whether the addition of Celebrex to EPO906 can reduce the incidence of grade 3-4 diarrhea to 6% or less. | Until 30 days after patient receives last study drug

SECONDARY OUTCOMES:
To estimate the time to progression, survival and response rate in patients with metastatic colorectal cancer who failed 5-FU/LV, CPT-11 and/or oxaliplatin based hemotherapy and receive Celebrex in combination with EPO906. | Until Patient goes off study
To further assess toxicity of this regimen. | 30 days after patient receives last dose
To investigate whether the molecular biomarkers including protein expression changes from plasma, the expression levels of VEGF, E-cadherin, TP, COX-2, and β-tubulin in tumor tissue associated with clinical outcome for this regimen. | Until Patient Death

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, M.D., Principal Investigator — U.S.C/Norris Cancer Center
Locations (1):
- U.S.C./Norris Comprehensive Cancer Center, Los Angeles, California, United States